CLINICAL TRIAL: NCT04149132
Title: Pulse Photoplethysmography as an Early Tool for the Diagnosis of Sepsis
Acronym: PROUD-1
Status: Completed | Type: Observational
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Other Study IDs: PROUD-1
Record Dates: First submitted 2019-10-29; First posted 2019-11-04 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Sepsis
Keywords: early diagnosis; infection; pulse photoplethysmography
MeSH Terms: conditions — Sepsis; Disease; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients without sepsis: Patients admitted and hospitalized for infections without sepsis and for other reasons in departments of Internal Medicine and Intensive Care Units
  Interventions: Device: pulse photoplethysmography (PPG); Diagnostic Test: Measurements of nitric oxide (NO) and malondialdehyde (MDA)

INTERVENTIONS:
Device: pulse photoplethysmography (PPG) — PPG and systolic blood pressure recording will be performed every two hours for three consecutive days. PPG reading will last two minutes and peaks of NO productions will be captured. Day 1 is considered the day of signing the informed consent followed by the first recording. On the first PPG recording of the same days i.e. on days 1, 2 and 3 the investigators will collect blood from the patients
Diagnostic Test: Measurements of nitric oxide (NO) and malondialdehyde (MDA) — On the first PPG recording of the same days i.e. on days 1, 2 and 3 the investigators will collect blood from the patients. NO will be measured in serum samples by the Griess reaction. MDA that is considered an index of oxidant status will be measured in serum samples by the thiobarbiturate assay and analysis by high-performance liquid chromatography (HPLC)

SUMMARY:
Early management of sepsis is associated with better outcome. However, this requires early recognition of the sepsis host. One recently developed customized pulse photoplethysmography (PPG) device manages to measure nitric oxide (NO) that is released from vascular endothelium and seems promising for earlier sepsis diagnosis than conventional approaches. Aim of the project To evaluate the diagnostic performance of the PPG device for the early diagnosis of sepsis is to evaluate the diagnostic performance of the PPG device for the early diagnosis of sepsis

DETAILED DESCRIPTION:
Sepsis is a life-threatening syndrome and the most common cause of death nowadays. This syndrome develops as a result of the dysregulated host response to an infectious insult. As such the mainstay of treatment is the early administration of antimicrobials leading to early eradication of the offending pathogen. However, in this statement the key-feature is the definition of what "early" means. Using the retrospective analysis of data associating final outcome from septic shock with the delay in start of antimicrobials from the start of vasopressors in 2713 patients with septic shock, it was found that 79.1% of patients in which this delay was less than one hour survived. Every further hour of delay in start of antibiotics led to 7.6% increase of the risk for unfavorable outcome. These findings were later confirmed from two other analyses. These findings generate two thoughts: a) the above results are based on early recognition of hospital-acquired sepsis that was achievable only because these studies were done in an Intensive Care Unit (ICU) environment in patients under close monitoring. However, early sepsis recognition for a newly admitted patient remains an unmet need; b) all the above results are coming from patients with septic shock where diagnosis had already been established since patients were already on vasopressors.

It is reasonable to hypothesize that if sepsis had been recognized even earlier final outcome would have been even better. Sanmina have developed a non-invasive technique for the measurement of endothelial released nitric oxide (NO) through customized pulse photoplethysmography (PPG). Since NO is released by the vascular endothelium early in the pathogenesis of sepsis it is reasonable to hypothesize that PPG is a technique that can early inform on the risk for a patient with suspicion of an infection to develop sepsis. The time of measurement is less than two minutes. Preliminary data show that the reading of a healthy subject of eight consecutive minutes cannot trace any increase of NO; in sepsis a peak of more than 200 units is shown within the first 40 seconds of measurement.

The development of PPG as a tool for the early diagnosis of sepsis requires a two-stage approach. The first stage is based on the association of PPG readings with the change of the SOFA (sequential organ failure assessment) score and vital signs to define if among patients who eventually develop sepsis, PPG changes will be produced earlier than changes of SOFA scores and of vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years
* Both genders
* Written informed consent provided by the patients or by first-degree relatives in case of patients unable to consent.
* Any of two:

Any infection in a patient with total SOFA score equal to 0 or 1 Patient without sepsis prone to the development of sepsis defined as patients with Charlson's Comorbidity Index (CCI) more than 2 irrespective the reason of admission. These patients are considered prone to infection based on previous findings of our group showing that CCI more than 2 is an independent predisposing factor for sepsis

Exclusion Criteria:

* Age below 18 years
* Denial to consent
* Any stage 4 malignancy
* Any do not resuscitate decision
* Active tuberculosis (TB) as defined by the co-administration of drugs for the treatment of TB
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Screening will be done for the inclusion and exclusion criteria in all patients admitted or hospitalized in the participating sites. Participants will be patients meeting all inclusion criteria and none of the exclusion criteria
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity of PPG for the diagnosis of sepsis. | 72 hours
  Sensitivity of PPG for the diagnosis of sepsis.

SECONDARY OUTCOMES:
Correlation of PPG (absolute number) with qSOFA score (absolute number) | 72 hours
  Correlation of PPG (absolute number) with qSOFA score (absolute number)
Correlation of PPG (absolute number) with SOFA score (absolute number) | 72 hours
  Correlation of PPG (absolute number) with SOFA score (absolute number)
Correlation of time (in minutes) of sepsis diagnosis between PPG (absolute number) and SOFA score (absolute number) | 72 hours
  Correlation of time (in minutes) of sepsis diagnosis between PPG (absolute number) and SOFA score (absolute number)
Correlation of time (in minutes) of sepsis diagnosis between PPG (absolute number) and hypotension (mmHg) | 72 hours
  Correlation of time (in minutes) of sepsis diagnosis between PPG (absolute number) and hypotension (mmHg)
The specificity, positive predictive value (PPV) and negative predictive value (NPV) of PPG for the diagnosis of sepsis | 72 hours
  The specificity, positive predictive value (PPV) and negative predictive value (NPV) of PPG for the diagnosis of sepsis
The sensitivity, specificity, PPV and NPV of PPG for the prognosis of 28-day outcome | 28 days
  The sensitivity, specificity, PPV and NPV of PPG for the prognosis of 28-day outcome
Correlation of PPG (absolute number) with circulating levels of NO (μmol/l) and MDA (μmol/l) | 72 hours
  The association between PPG and circulating levels of NO and MDA

CONTACTS AND LOCATIONS:
Overall Officials: Antonios Papadopoulos, MD, PhD, Principal Investigator — 4th Department of Internal Medicine
Locations (4):
- Greece (4):
  - Intensive Care Unit, "Korgialenio - Benakio" General Hospital of Athens, Athens
  - Department of Clinical Therapeutics, "Alexandra" General Hospital of Athens, National and Kapodistrian University of Athens, Medical School, Athens
  - 2nd Department of Critical Care, "Attikon" University Hospital, National and Kapodistrian University of Athens, Medical School, Athens
  - 4th Department of Internal Medicine, "Attikon" University Hospital, National and Kapodistrian University of Athens, Medical School, Athens

IPD SHARING:
Plan to Share IPD: Undecided